CLINICAL TRIAL: NCT01475682
Title: Long Term Cardiovascular Complications in Men With Obstructive Sleep Apnea - Prospective 9 Years Follow-up Study
Brief Title: Long Term Cardiovascular Complications in Men With Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lam Jamie Chung Mei, Honorary Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW 10-002
Record Dates: First submitted 2011-11-16; First posted 2011-11-21 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Obstructive Sleep Apnea; Cardiovascular Diseases; Metabolic Diseases
Keywords: Obstructive sleep apnea; cardiometabolic complications; Effects of CPAP treatment
MeSH Terms: conditions — Sleep Apnea, Obstructive; Cardiovascular Diseases; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: 167 subjects recruited from our previous "OSA and metabolic syndrome" (OSAMS) cohort from October 2002 to June 2007 will be invited to be reassessed at this time point.

SUMMARY:
Subjects with Obstructive Sleep Apnea (OSA) are at increased risk of developing cardiometabolic complications, and effective long-term nCPAP treatment significantly reduces the risk of cardiovascular morbidity and mortality.

DETAILED DESCRIPTION:
1. Primary outcome:

   Incidence of cardiometabolic diseases in subjects with OSA over 9 years.
2. Secondary outcomes:

Effects of CPAP treatment on cardiometabolic conditions

ELIGIBILITY:
Inclusion Criteria:

* From previous cohort for reassessment.

Exclusion Criteria:

* Unstable medical conditions

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 167 subjects recruited from our previous "OSA and metabolic syndrome" (OSAMS) cohort from October 2002 to June 2007 will be invited to be reassessed at this time point.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Estimated)
Dates: Start 2011-11; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiometabolic complications | 9 years
  167 subjects recruited from our previous "OSA and metabolic syndrome" (OSAMS) cohort from October 2002 to June 2007 will be invited to be reassessed at this time point.

SECONDARY OUTCOMES:
Effects of CPAP treatment on cardiometabolic conditions | 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Jamie C Lam, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong